CLINICAL TRIAL: NCT00638066
Title: Comparison of Efficacy of 250 Units Versus 500 Units of Botulinum Toxin in the Treatment of Refractory Vaginismus
Brief Title: Botulinum Toxin Injection for Treatment of Vaginismus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Dr Shirin Ghazizadeh, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 130/6/6081; 130/6/6081
Record Dates: First submitted 2008-01-10; First posted 2008-03-18 (Estimated); Last update posted 2008-03-18 (Estimated); Status verified 2008-03

CONDITIONS: Vaginismus
Keywords: vaginismus; botulinum toxin A; dyspareunia; unconsummated marriage
MeSH Terms: conditions — Vaginismus; Dyspareunia | interventions — Botulinum Toxins; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: botulinum toxin A
- 2 (Active Comparator)
  Interventions: Drug: botulinum toxin

INTERVENTIONS:
Drug: botulinum toxin — 500 units of botulinum toxin for the second arm
  Arms: 2
Drug: botulinum toxin A — 250 units of botulinum toxin A once
  Arms: 1

SUMMARY:
According to high rate of vaginismus (about 10 percent) which leads to unconsummated marriage (about 1 percent) and low efficacy for conventional treatments such as biofeedback therapy, analgesic drugs and pain killers and surgical treatment, there's necessity to find more effective method.

In our previous study, injecting botulinum toxin in 23 patients cured 75% of them.Now we are to make comparison between different doses of toxin injection and record the patient sexual satisfaction.

DETAILED DESCRIPTION:
Vaginismus is the recurrent or persistent involuntary contraction of the perineal muscles surrounding the outer third of the vagina when penile, finger, tampon, or speculum penetration is attempted . Vaginismus can be primary, in which the women has never been able to have intercourse, or secondary, which is often due to acquired dyspareunia. It is relatively rare, affecting about 1% of women . Treatment of vaginismus is directed toward extinguishing the conditioned involuntary vaginal spasm. This can be accomplished by teaching Kegel exercises to acquaint the patient with voluntary control of her levator muscles. Medications such as lubricants, anesthetic creams, propranolol, or alprazolam to reduce anxiety have been used effectively, but approximately 10% of patients do not respond. Botulinum toxin type A has been successfully used to treat a wide range of muscular disorders such as strabismus, blepharospasm, and cervical dystonia. It is also been used to reduce facial lines and wrinkles.The extent of paralysis depends on the amount of toxin to which there is exposure relative to muscle bulk.In our previous study, one week after injecting botulinum toxin in 23 patients (95.8%) had a vaginal exam, which showed no or little resistance; 18 (75%) achieved satisfactory intercourse after the first injection. Now we are to make comparison between different doses of toxin injection and record the patient sexual satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Unconsummated marriage
* Difficult mating
* No response to biofeedback

Exclusion Criteria:

* Patient unlikely to have toxin injection
* Not having mutual life with partner
* Non treated pelvic and vaginal infection

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-04 (Estimated); Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
50 percent of patient satisfaction | first two month

SECONDARY OUTCOMES:
total patient satisfaction | next four month

CONTACTS AND LOCATIONS:
Overall Officials: Abbas noroozi, PhD, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Tehran University of Medical Sciences, Vali e Asr Reproductive Health Research Center, Tehran, Tehran Province, Iran